CLINICAL TRIAL: NCT02197572
Title: A Phase 1 Study to Evaluate the Effect of MLN0128 on the QTc Interval in Patients With Advanced Solid Tumors
Brief Title: Effect of Sapanisertib (MLN0128) on the QTc Interval in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C31002; U1111-1156-4099 (Other: World Health Organization)
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Advanced Solid Tumors
Keywords: Drug therapy
MeSH Terms: interventions — sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sapanisertib (Experimental): Sapanisertib starting dose of 40 mg, capsules, orally, once, on Day 1, Cycle 1 (28 days cycle) followed by sapanisertib 30 mg, capsules, orally, once weekly (QW) starting on Cycle 1, Day 8 based on safety and tolerability and as per investigator's discretion up to disease progression, unacceptable sapanisertib-related toxicity, withdrawal of consent, or for up to 12 months (whichever occurred first).
  Interventions: Drug: Sapanisertib

INTERVENTIONS:
Drug: Sapanisertib — Sapanisertib capsules.
  Other Names: MLN0128; INK128; TAK-228

SUMMARY:
The purpose of this study is to characterize the effect of a single dose of 40 mg sapanisertib (MLN0128) on the electrocardiographic QT/QTc interval in participants with advanced solid tumors.

DETAILED DESCRIPTION:
The drug being tested in this study is called sapanisertib (MLN0128). Sapanisertib is being tested to determine the effect of a single 40 mg dose on the electrocardiographic measure of the time between the start of the Q wave and the end of the T wave in the electrical cycle of the heart (QT)/rate corrected QT (QTc) interval in patients with advanced solid tumors. This study will look at electrocardiogram (ECG) results before and after a single dose of sapanisertib.

The study will enroll approximately 30 patients. All participants will receive a single 40 mg dose of sapanisertib capsules on Day 1. Participants may continue to receive sapanisertib for up to 1 year at a dose of up to 30 mg once weekly if a clinical benefit is being derived.

This multi-centre trial will be conducted in the United States. The overall time to participate in this study is up to 14 months. Participants will make 6 visits to the clinic and end of study visit 30 to 40 days after last dose of study drug for a follow-up assessment. Participants that continue treatment with sapanisertib will continue to make additional visits to the clinic once or twice every 4 weeks and the end of study visit 30 to 40 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria

* Men or women participants 18 years or older.
* Must have a radiographically or clinically evaluable solid tumor Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Female participants who are postmenopausal for at least 1 year before the screening visit, OR are surgically sterile, OR if they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 3 months after the last dose of study drug, OR agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Male participants, even if surgically sterilized (i.e., status post vasectomy), who agree to practice effective barrier contraception during the entire study treatment period and through 3 months after the last dose of study drug, or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.)
* Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
* Ability to swallow oral medications, willingness to perform mucositis prophylaxis, and suitable venous access for the study-required blood sampling.

Exclusion Criteria

* Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the screening period.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Treatment with any investigational products within 14 days before the first dose of study drug and systemic anticancer therapy within 28 days before the first dose of study drug.
* Untreated brain metastasis or history of leptomeningeal disease or spinal cord compression.
* Tumors with involvement of the mediastinum.
* Failure to recover from the reversible effects of prior anticancer therapies with the exception of alopecia, and after-effects associated with prior tyrosine kinase inhibitor therapy such as hair depigmentation, hypothyroidism, and/or splinter hemorrhage.
* Systemic corticosteroid (inhalers are allowed) within 7 days before the first dose of study drug.
* Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown or other reason that may alter the absorption of Sapanisertib.
* Diagnosis of diabetes mellitus; participants with a history of transient glucose intolerance due to corticosteroid administration may be enrolled if all other inclusion/exclusion criteria are met.
* Significant active cardiovascular or pulmonary disease at study entry
* History of arrhythmia requiring an implantable cardiac defibrillator
* Clinically significant comorbidities such as uncontrolled pulmonary disease, active central nervous system disease, active infection, serious infection within 14 days before the first dose of study drug, or any other condition that could compromise study participation by the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - Sarasota, Florida
  - St Louis, Missouri
  - The Bronx, New York
  - Oklahoma City, Oklahoma
  - Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Patel C, Goel S, Patel MR, Rangachari L, Wilbur JD, Shou Y, Venkatakrishnan K, Lockhart AC. Phase 1 Study to Evaluate the Effect of the Investigational Anticancer Agent Sapanisertib on the QTc Interval in Patients With Advanced Solid Tumors. Clin Pharmacol Drug Dev. 2020 Oct;9(7):876-888. doi: 10.1002/cpdd.808. Epub 2020 Jun 2. PMID 32488989

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in the United States from 15 Sep 2014 to 28 Feb 2019.
Pre-assignment Details: Participants who had advanced solid tumors were enrolled to receive sapanisertib 40 mg on Day 1. Participants then received sapanisertib 30 mg once weekly (QW) until they experienced disease progression or unacceptable sapanisertib-related toxicity or withdrawal of consent or for up to 12 months (whichever occurred first).
Period: Overall Study
Arm/Group | Sapanisertib
Started | 44
Completed | 0
Not Completed | 44
Not completed — Progressive Disease | 28
Not completed — Withdrawal by Subject | 9
Not completed — Adverse Event | 3
Not completed — Reason Not Specified | 4

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of Sapanisertib.
Groups:
- Sapanisertib: Sapanisertib starting dose of 40 mg, capsules, orally, once, on Day 1, Cycle 1 followed by sapanisertib 30 mg, capsules, orally, once weekly (QW) starting on Cycle 1, Day 8 based on safety and tolerability and as per investigator's discretion up to disease progression, unacceptable sapanisertib-related toxicity, withdrawal of consent, or for up to 12 months (whichever occurred first).
Arm/Group | Sapanisertib
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 30
  More than one race | 0
  Unknown or Not Reported | 5
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is the number of participants with evaluable data at Baseline.
  cm
    number analyzed (Participants) | 42
    (all) | 166.8 (8.61)
Weight [Mean (Standard Deviation); unit: kg] | 74.9 (16.08)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=weight(kg)/height(m)^2 Population: Number analyzed is the number of participants with evaluable data at Baseline.
  kg/m^2
    number analyzed (Participants) | 42
    (all) | 27.141 (5.8591)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Time-Matched Baseline in QTcI, Individual Baseline Corrected Rate-Corrected QT Interval
Description: The mean changes of QTcI from time-matched baseline was measured by electrocardiogram (ECG) to evaluate the potential effect of drug on QTc interval duration. Holter monitors were used to collect triplicate ECG measurements and were based on a repeated measures mixed effects linear model. A negative change from baseline indicates shortening and a positive change from baseline indicates prolongation of QTcI interval.
Time Frame: Baseline; Cycle 1 (28 days cycle): 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 24 and 48 hours postdose
Population: Primary analysis population: participants that have all timepoints collected on Holter ECG monitoring on Day -1 and Day 1 of Cycle 1 including ECG timepoints on Cycle 1 Days 1 to 3 at 24 or 48 hours postdose and baseline comparisons available for these analyses. Number analyzed is number of participants with evaluable data at given time-point.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Sapanisertib
Number analyzed (Participants) | 32
msec
  Change from Baseline at 0.25 Hours Postdose: number analyzed (Participants) | 28
  Change from Baseline at 0.25 Hours Postdose | -1.3 (9.5)
  Change from Baseline at 0.5 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 0.5 Hours Postdose | -7.7 (9.8)
  Change from Baseline at 1 Hour Postdose: number analyzed (Participants) | 30
  Change from Baseline at 1 Hour Postdose | -1.1 (11.5)
  Change from Baseline at 1.5 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 1.5 Hours Postdose | -2.0 (12.5)
  Change from Baseline at 2 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 2 Hours Postdose | -4.2 (11.2)
  Change from Baseline at 2.5 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 2.5 Hours Postdose | -6.9 (10.6)
  Change from Baseline at 3 Hours Postdose: number analyzed (Participants) | 28
  Change from Baseline at 3 Hours Postdose | -8.5 (11.2)
  Change from Baseline at 4 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 4 Hours Postdose | -6.6 (9.3)
  Change from Baseline at 6 Hours Postdose | -8.8 (15.6)
  Change from Baseline at 8 Hours Postdose: number analyzed (Participants) | 27
  Change from Baseline at 8 Hours Postdose | -1.3 (14.1)
  Change from Baseline at 10 Hours Postdose: number analyzed (Participants) | 13
  Change from Baseline at 10 Hours Postdose | -5.6 (17.5)
  Change from Baseline at 24 Hours Postdose | 7.1 (25.4)
  Change from Baseline at 48 Hours Postdose: number analyzed (Participants) | 19
  Change from Baseline at 48 Hours Postdose | 3.1 (17.8)
Statistical Analysis 1: Comparison: Sapanisertib; Change from Baseline at 0.25 Hours Postdose; Test type: Other; Least Squares Mean = -2.2, 95% CI 1-sided [upper limit 2.2]
Statistical Analysis 2: Comparison: Sapanisertib; Change from Baseline at 0.5 Hours Postdose; Test type: Other; Least Squares Mean = -8.3, 95% CI 1-sided [upper limit -4.0]
Statistical Analysis 3: Comparison: Sapanisertib; Change from Baseline at 1 Hour Postdose; Test type: Other; Least Squares Mean = -1.8, 95% CI 1-sided [upper limit 2.6]
Statistical Analysis 4: Comparison: Sapanisertib; Change from Baseline at 1.5 Hours Postdose; Test type: Other; Least Squares Mean = -2.7, 95% CI 1-sided [upper limit 1.7]
Statistical Analysis 5: Comparison: Sapanisertib; Change from Baseline at 2 Hours Postdose; Test type: Other; Least Squares Mean = -5.0, 95% CI 1-sided [upper limit -0.6]
Statistical Analysis 6: Comparison: Sapanisertib; Change from Baseline at 2.5 Hours Postdose; Test type: Other; Least Squares Mean = -7.6, 95% CI 1-sided [upper limit -3.2]
Statistical Analysis 7: Comparison: Sapanisertib; Change from Baseline at 3 Hours Postdose; Test type: Other; Least Squares Mean = -9.1, 95% CI 1-sided [upper limit -4.6]
Statistical Analysis 8: Comparison: Sapanisertib; Change from Baseline at 4 Hours Postdose; Test type: Other; Least Squares Mean = -7.2, 95% CI 1-sided [upper limit -2.9]
Statistical Analysis 9: Comparison: Sapanisertib; Change from Baseline at 6 Hours Postdose; Test type: Other; Least Squares Mean = -8.8, 95% CI 1-sided [upper limit -4.6]
Statistical Analysis 10: Comparison: Sapanisertib; Change from Baseline at 8 Hours Postdose; Test type: Other; Least Squares Mean = -2.2, 95% CI 1-sided [upper limit 2.4]
Statistical Analysis 11: Comparison: Sapanisertib; Change from Baseline at 10 Hours Postdose; Test type: Other; Least Squares Mean = -6.6, 95% CI 1-sided [upper limit -0.5]
Statistical Analysis 12: Comparison: Sapanisertib; Change from Baseline at 24 Hours Postdose; Test type: Other; Least Squares Mean = 7.1, 95% CI 1-sided [upper limit 11.4]
Statistical Analysis 13: Comparison: Sapanisertib; Change from Baseline at 48 Hours Postdose; Test type: Other; Least Squares Mean = 2.8, 95% CI 1-sided [upper limit 8.1]

2. Secondary Outcome: Number of Participants With Atleast One Adverse Event (AE) and Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. An SAE is any untoward medical occurrence that results in death; is life-threatening; requires inpatient hospitalization or prolongation of present hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect or is a medically important event that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the participant or may require intervention to prevent one of other outcomes listed in definition above, or involves suspected transmission via a medicinal product of an infectious agent.
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (Up to 13 months)
Population: Safety population included all participants who received at least 1 dose of sapanisertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Sapanisertib
Number analyzed (Participants) | 44
Participants
  AE | 43
  SAE | 18

3. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Laboratory Values Reported as AE
Description: The laboratory parameters included clinical chemistry, hematology, and urinalysis. Any abnormal change in the laboratory values were assessed by Investigator and reported as AE. An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (Up to 13 months)
Population: Safety population included all participants who received at least 1 dose of sapanisertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Sapanisertib
Number analyzed (Participants) | 44
Participants
  Blood Creatinine Increased | 2
  Blood Triglycerides Increased | 2
  Hyperglycemia | 8
  Hypertriglyceridemia | 1
  Hypomagnesemia | 1
  Hypophosphatemia | 2
  Vitamin D Deficiency | 2
  Anemia | 3
  Thrombocytopenia | 1

4. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Vital Signs Reported as AE
Description: Vital sign measurements included blood pressure (diastolic and systolic), heart rate, and temperature. Any abnormal change in the vital sign values were assessed by Investigator and reported as AE. An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (Up to 13 months)
Population: Safety population included all participants who received at least 1 dose of sapanisertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Sapanisertib
Number analyzed (Participants) | 44
Participants
  Hypotension | 1
  Postoperative Fever | 1
  Pyrexia | 4

5. Secondary Outcome: Mean Change From Time-Matched Baseline in QTc With Rate-Corrected QT Interval With Bazett Correction (QTcB)
Description: The mean changes of QTcB from time-matched baseline was measured by ECG to evaluate the potential effect of drug on QTc interval duration. Holter monitors were used to collect triplicate ECG measurements and were based on a repeated measures mixed effects linear model. A negative change from baseline indicates shortening and a positive change from baseline indicates prolongation of QTcB interval.
Time Frame: Baseline; Cycle 1 (28 days cycle): 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 24 and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Sapanisertib
Number analyzed (Participants) | 32
msec
  Change from Baseline at 0.25 Hours Postdose: number analyzed (Participants) | 28
  Change from Baseline at 0.25 Hours Postdose | -1.9 (9.7)
  Change from Baseline at 0.5 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 0.5 Hours Postdose | -9.8 (12.1)
  Change from Baseline at 1 Hour Postdose: number analyzed (Participants) | 30
  Change from Baseline at 1 Hour Postdose | -2.0 (12.4)
  Change from Baseline at 1.5 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 1.5 Hours Postdose | -3.1 (13.5)
  Change from Baseline at 2 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 2 Hours Postdose | -5.1 (11.4)
  Change from Baseline at 2.5 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 2.5 Hours Postdose | -7.5 (10.6)
  Change from Baseline at 3 Hours Postdose: number analyzed (Participants) | 28
  Change from Baseline at 3 Hours Postdose | -8.3 (14.6)
  Change from Baseline at 4 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 4 Hours Postdose | -8.5 (8.7)
  Change from Baseline at 6 Hours Postdose | -5.9 (12.2)
  Change from Baseline at 8 Hours Postdosen: number analyzed (Participants) | 27
  Change from Baseline at 8 Hours Postdosen | 1.9 (13.7)
  Change from Baseline at 10 Hours Postdose: number analyzed (Participants) | 13
  Change from Baseline at 10 Hours Postdose | -4.4 (15.3)
  Change from Baseline at 24 Hours Postdose | 11.9 (17.0)
  Change from Baseline at 48 Hours Postdose: number analyzed (Participants) | 19
  Change from Baseline at 48 Hours Postdose | 7.6 (14.9)

6. Secondary Outcome: Mean Change From Time-Matched Baseline in QTc With Rate-Corrected QT Interval Fridericia Correction (QTcF)
Description: The mean changes of QTcF from time-matched baseline was measured by ECG to evaluate the potential effect of drug on QTc interval duration. Holter monitors were used to collect triplicate ECG measurements and were based on a repeated measures mixed effects linear model. A negative change from baseline indicates shortening and a positive change from baseline indicates prolongation of QTcF interval.
Time Frame: Baseline; Cycle 1 (28 days cycle): 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 24 and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Sapanisertib
Number analyzed (Participants) | 32
msec
  Change from Baseline at 0.25 Hours Postdose: number analyzed (Participants) | 28
  Change from Baseline at 0.25 Hours Postdose | -1.3 (8.5)
  Change from Baseline at 0.5 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 0.5 Hours Postdose | -5.0 (10.6)
  Change from Baseline at 1 Hour Postdose: number analyzed (Participants) | 30
  Change from Baseline at 1 Hour Postdose | 2.1 (12.0)
  Change from Baseline at 1.5 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 1.5 Hours Postdose | 0.6 (12.7)
  Change from Baseline at 2 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 2 Hours Postdose | -3.3 (12.2)
  Change from Baseline at 2.5 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 2.5 Hours Postdose | -7.0 (11.1)
  Change from Baseline at 3 Hours Postdose: number analyzed (Participants) | 28
  Change from Baseline at 3 Hours Postdose | -7.4 (13.2)
  Change from Baseline at 4 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 4 Hours Postdose | -7.7 (10.3)
  Change from Baseline at 6 Hours Postdose | -10.1 (13.0)
  Change from Baseline at 8 Hours Postdose: number analyzed (Participants) | 27
  Change from Baseline at 8 Hours Postdose | -4.0 (15.1)
  Change from Baseline at 10 Hours Postdose: number analyzed (Participants) | 13
  Change from Baseline at 10 Hours Postdose | -11.9 (16.1)
  Change from Baseline at 24 Hours Postdose | 0.8 (16.0)
  Change from Baseline at 48 Hours Postdose: number analyzed (Participants) | 19
  Change from Baseline at 48 Hours Postdose | 2.5 (13.2)

7. Secondary Outcome: Change From Time-Matched Baseline in QRS Interval
Description: QRS interval is defined as the time between the start of the Q wave and end of the S wave on ECG. Holter monitors were used to collect triplicate ECG measurements and were based on a repeated measures mixed effects linear model. A negative change from baseline indicates shortening and a positive change from baseline indicates prolongation of QRS interval.
Time Frame: Baseline; Cycle 1 (28 days cycle): 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 24 and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Sapanisertib
Number analyzed (Participants) | 32
msec
  Change from Baseline at 0.25 Hours Postdose: number analyzed (Participants) | 28
  Change from Baseline at 0.25 Hours Postdose | -0.7 (3.3)
  Change from Baseline at 0.5 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 0.5 Hours Postdose | -1.4 (3.3)
  Change from Baseline at 1 Hour Postdose: number analyzed (Participants) | 30
  Change from Baseline at 1 Hour Postdose | -2.8 (2.9)
  Change from Baseline at 1.5 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 1.5 Hours Postdose | -1.8 (4.1)
  Change from Baseline at 2 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 2 Hours Postdose | -1.4 (4.0)
  Change from Baseline at 2.5 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 2.5 Hours Postdose | -2.3 (4.7)
  Change from Baseline at 3 Hours Postdose: number analyzed (Participants) | 28
  Change from Baseline at 3 Hours Postdose | -2.4 (3.2)
  Change from Baseline at 4 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 4 Hours Postdose | -2.9 (3.2)
  Change from Baseline at 6 Hours Postdose | -1.3 (3.0)
  Change from Baseline at 8 Hours Postdosen: number analyzed (Participants) | 27
  Change from Baseline at 8 Hours Postdosen | -0.8 (4.1)
  Change from Baseline at 10 Hours Postdose: number analyzed (Participants) | 13
  Change from Baseline at 10 Hours Postdose | -4.0 (6.5)
  Change from Baseline at 24 Hours Postdose | -1.4 (4.0)
  Change from Baseline at 48 Hours Postdose: number analyzed (Participants) | 19
  Change from Baseline at 48 Hours Postdose | 0.2 (5.3)

8. Secondary Outcome: Change From Time-Matched Baseline in PR Interval
Description: PR interval is defined as the time between the start of the P wave and the beginning of the QRS complex on ECG. Holter monitors were used to collect triplicate ECG measurements and were based on a repeated measures mixed effects linear model. A negative change from baseline indicates shortening and a positive change from baseline indicates prolongation of PR interval.
Time Frame: Baseline; Cycle 1 (28 days cycle): 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 24 and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Sapanisertib
Number analyzed (Participants) | 32
msec
  Change from Baseline at 0.25 Hours Postdose: number analyzed (Participants) | 28
  Change from Baseline at 0.25 Hours Postdose | -1.8 (13.9)
  Change from Baseline at 0.5 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 0.5 Hours Postdose | -0.8 (13.6)
  Change from Baseline at 1 Hour Postdose: number analyzed (Participants) | 30
  Change from Baseline at 1 Hour Postdose | 0.7 (11.5)
  Change from Baseline at 1.5 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 1.5 Hours Postdose | -0.7 (11.4)
  Change from Baseline at 2 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 2 Hours Postdose | -1.7 (9.3)
  Change from Baseline at 2.5 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 2.5 Hours Postdose | 0.1 (11.7)
  Change from Baseline at 3 Hours Postdose: number analyzed (Participants) | 28
  Change from Baseline at 3 Hours Postdose | -2.7 (10.8)
  Change from Baseline at 4 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 4 Hours Postdose | -1.9 (13.3)
  Change from Baseline at 6 Hours Postdose | -8.9 (13.2)
  Change from Baseline at 8 Hours Postdosen: number analyzed (Participants) | 27
  Change from Baseline at 8 Hours Postdosen | -7.3 (11.4)
  Change from Baseline at 10 Hours Postdose: number analyzed (Participants) | 13
  Change from Baseline at 10 Hours Postdose | -12.3 (11.5)
  Change from Baseline at 24 Hours Postdose | -6.8 (15.7)
  Change from Baseline at 48 Hours Postdose: number analyzed (Participants) | 19
  Change from Baseline at 48 Hours Postdose | -2.9 (20.7)

9. Secondary Outcome: Change From Time-Matched Baseline in Heart Rate
Description: Heart rate was assessed using the ECG. Holter monitors were used to collect triplicate ECG measurements and were based on a repeated measure mixed effects linear model. A negative change from baseline indicates decrease in heart rate.
Time Frame: Baseline; Cycle 1 (28 days cycle): 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 24 and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Sapanisertib
Number analyzed (Participants) | 32
beats per minute (bpm)
  Change from Baseline at 0.25 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 0.25 Hours Postdose | -0.9 (5.7)
  Change from Baseline at 0.5 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 0.5 Hours Postdose | -4.7 (5.9)
  Change from Baseline at 1 Hour Postdose: number analyzed (Participants) | 30
  Change from Baseline at 1 Hour Postdose | -4.2 (6.6)
  Change from Baseline at 1.5 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 1.5 Hours Postdose | -3.7 (6.0)
  Change from Baseline at 2 Hours Postdose: number analyzed (Participants) | 31
  Change from Baseline at 2 Hours Postdose | -1.0 (8.2)
  Change from Baseline at 2.5 Hours Postdose: number analyzed (Participants) | 30
  Change from Baseline at 2.5 Hours Postdose | -0.3 (4.8)
  Change from Baseline at 3 Hours Postdose: number analyzed (Participants) | 31
  Change from Baseline at 3 Hours Postdose | -0.3 (7.2)
  Change from Baseline at 4 Hours Postdose: number analyzed (Participants) | 31
  Change from Baseline at 4 Hours Postdose | -0.4 (10.1)
  Change from Baseline at 6 Hours Postdose | 4.8 (6.3)
  Change from Baseline at 8 Hours Postdose: number analyzed (Participants) | 29
  Change from Baseline at 8 Hours Postdose | 7.0 (9.7)
  Change from Baseline at 10 Hours Postdose: number analyzed (Participants) | 13
  Change from Baseline at 10 Hours Postdose | 7.9 (9.2)
  Change from Baseline at 24 Hours Postdose | 12.4 (11.8)
  Change from Baseline at 48 Hours Postdose: number analyzed (Participants) | 20
  Change from Baseline at 48 Hours Postdose | 5.0 (9.8)

10. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Sapanisertib
Time Frame: Cycle 1 (28 days cycle), Day 1, predose and at multiple timepoints (Up to 48 hours) postdose
Population: Pharmacokinetic (PK) analysis population included all participants who received at least 1 dose of sapanisertib and had sufficient concentration-time data to calculate 1 or more PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sapanisertib
Number analyzed (Participants) | 44
ng/mL | 337.1 (178.27)

11. Secondary Outcome: Tmax: Time to Reach Cmax for Sapanisertib
Time Frame: Cycle 1 (28 days cycle), Day 1, predose and at multiple timepoints (Up to 48 hours) postdose
Population: PK analysis population included all participants who received at least 1 dose of sapanisertib and had sufficient concentration-time data to calculate 1 or more PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Sapanisertib
Number analyzed (Participants) | 44
hours | 1.5167 [0.500 to 24.000]

12. Secondary Outcome: AUCt: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of Last Measurable Concentration for Sapanisertib
Time Frame: Cycle 1 (28 days cycle), Day 1, predose and at multiple timepoints (Up to 48 hours) postdose
Population: PK analysis population included all participants who received at least 1 dose of sapanisertib and had sufficient concentration-time data to calculate 1 or more PK parameters. Overall number of participants analyzed were participants with data available for analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Sapanisertib
Number analyzed (Participants) | 37
h*ng/mL | 2875.7406 (2110.90918)

13. Secondary Outcome: AUCinf: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for Sapanisertib
Time Frame: Cycle 1 (28 days cycle), Day 1, predose and at multiple timepoints (Up to 48 hours) postdose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Sapanisertib
Number analyzed (Participants) | 36
h*ng/mL | 2992.5394 (2405.41705)

14. Secondary Outcome: T1/2: Terminal Elimination Half-life for Sapanisertib
Time Frame: Cycle 1 (28 days cycle), Day 1, predose and at multiple timepoints (Up to 48 hours) postdose
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | Sapanisertib
Number analyzed (Participants) | 36
hours | 9.0682 [4.477 to 16.867]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (Up to 13 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Sapanisertib
All-Cause Mortality (participants affected / at risk) | 2/44
Serious Adverse Events (participants affected / at risk) | 18/44
Other Adverse Events (participants affected / at risk) | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sapanisertib (N=44)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Small Intestinal Perforation (Gastrointestinal disorders) | 1 — One treatment-emergent death occurred during treatment with sapanisertib and is not related.
Stomatitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Bile Duct Obstruction (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Appendicitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Post Procedural Fever (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — One treatment-emergent death occurred during treatment with sapanisertib and is not related.
Mental Status Changes (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sapanisertib (N=44)
Anaemia (Blood and lymphatic system disorders) | 3
Sinus Tachycardia (Cardiac disorders) | 4
Vision Blurred (Eye disorders) | 5
Nausea (Gastrointestinal disorders) | 35
Vomiting (Gastrointestinal disorders) | 25
Diarrhoea (Gastrointestinal disorders) | 15
Stomatitis (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 9
Dry Mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 5
Abdominal Pain (Gastrointestinal disorders) | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 28
Chills (General disorders) | 4
Gait Disturbance (General disorders) | 4
Pyrexia (General disorders) | 4
Oedema Peripheral (General disorders) | 3
Urinary Tract Infection (Infections and infestations) | 13
Fall (Injury, poisoning and procedural complications) | 4
Weight Decreased (Investigations) | 14
Decreased Appetite (Metabolism and nutrition disorders) | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 9
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 9
Headache (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 3
Depression (Psychiatric disorders) | 6
Anxiety (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 5
Dysuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT02197572/Prot_000.pdf
  • Statistical Analysis Plan (2015-02-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT02197572/SAP_001.pdf